CLINICAL TRIAL: NCT01683747
Title: Single Dose Enteral Tranexamic Acid for the Reduction of Morbidity in Hospitalized Critically Ill Patients
Brief Title: Single Dose Enteral Tranexamic Acid in Critically Ill Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lower than anticipated enrollment
Sponsor: San Diego Veterans Healthcare System (U.S. Federal Agency)
Collaborators: Inflammagen/Leading Ventures (Unknown)
Responsible Party: Principal Investigator, Erik B. Kistler, MD, PhD, Principal Investigator, Assistant Professor, San Diego Veterans Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 110376
Record Dates: First submitted 2012-09-09; First posted 2012-09-12 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Shock; Sepsis; Hypotension; Critical Illness
Keywords: sepsis; shock; placebo controlled; double blinded; interventional
MeSH Terms: conditions — Shock; Sepsis; Hypotension; Critical Illness | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic acid (Experimental): Study group receives enteral tranexamic acid in normal saline in addition to usual care.
  Interventions: Drug: Tranexamic Acid
- Control group (Placebo Comparator): Control group receives vehicle (normal saline) without study drug and usual care.
  Interventions: Drug: Control Intervention (Carrier fluid only)

INTERVENTIONS:
Drug: Tranexamic Acid
  Other Names: Cyclokapron
  Arms: Tranexamic acid
Drug: Control Intervention (Carrier fluid only)
  Arms: Control group

SUMMARY:
The premise of this study is that enteral tranexamic acid will help to maintain small bowel integrity, which is often compromised by critical illness due to inadequate cardiovascular perfusion (i.e., shock), and that maintenance of small bowel integrity will decrease morbidity in critically ill patients.

DETAILED DESCRIPTION:
The primary objective of this study is to provide preliminary efficacy and safety data on the enteral administration of a one-time dose of tranexamic acid to critically ill patients for the reduction of morbidity at 28 days after enrollment in the study.

Secondary objectives of this study are to determine the efficacy of administration of enteral tranexamic acid in reducing intensive care unit (ICU) and hospital length-of-stay, as well and mortality and morbidity at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients admitted to ICU within 48 hours of onset of illness
* Patients with feeding tubes (e.g., orogastric, nasogastric, PEG, etc.)

Exclusion Criteria:

* primary admitting diagnosis of cancer
* primary admitting diagnosis of acute congestive heart failure
* primary admitting diagnosis of chronic obstructive pulmonary disease (COPD)
* primary admitting diagnosis of acute myocardial infarction or unstable cardiac arrythmia
* primary admitting diagnosis of amyotrophic lateral sclerosis (ALS) or other non-infectious disease
* primary admitting diagnosis of post-operative neurosurgical procedure
* known hypersensitivity to tranexamic acid
* acquired disturbances of color vision
* hematuria cause by disease of the renal parenchyma
* active thromboembolic disease such as deep venous thrombosis or pulmonary embolism
* patients with known clotting disorders or other known bleeding disorders
* recent (within 3 months) or active cerebrovascular bleed
* pregnancy
* inability to take study medicine (i.e., ileus with > 500ml stomach residuals, NPO status)
* patients excluded at the discretion of the treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Morbidity | 28 days
  Morbidity will be assessed at 28 days as measured by the validated Self-Administered Quality of Well-being Scale (QWB-SA) and 5-Point modified Oxford Handicap Scale [secondary scale]

SECONDARY OUTCOMES:
morbidity | 6 months
  Morbidity will be assessed at 28 days as measured by the validated Self-Administered Quality of Well-being Scale (QWB-SA) and 5-Point modified Oxford Handicap Scale [secondary scale]
mortality | 28 days
  All-cause death will be measured at 28 days
mortality | 6 months
  All cause mortality will be measured at 6 months
ICU length of stay | up to 6 months
  Time spent as a patient in the ICU will be measured
Hospital length of stay | up to 6 months
  Time spent in the hospital as a patient will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Erik B Kistler, MD, PhD, Principal Investigator — VA San Diego Healthcare/University of California, San Diego
Locations (1):
- VA San Diego Health Care System, San Diego, California, United States